CLINICAL TRIAL: NCT01936220
Title: Relapse Prevention in First Episode of Schizophrenia and Related Psychotic Disorders: a 5 Year Randomized Controlled Trial
Brief Title: Relapse Prevention in First Episode Schizophrenia: a 5 Year Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Donald H. Linszen, Principle Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Grant 28-1241-2
Record Dates: First submitted 2013-08-23; First posted 2013-09-06 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; First-psychotic episode; Initial phase; Relapse prevention; Specialized treatment; Parent groups; Social functioning
MeSH Terms: conditions — Schizophrenia; Social Adjustment | interventions — Secondary Prevention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Continuity of specialized care (Experimental): Continuity of specialized inpatient and outpatient care (relapse prevention)
  Interventions: Behavioral: Continuity of specialized care
- Continuity of specialized care and parent groups (Experimental): Continuity of specialized care combined with Parent groups
  Interventions: Behavioral: Continuity of specialized care; Behavioral: Parent groups combined with Continuity of Specialized care
- Treatment as usual (Active Comparator): Discontinuity of care, relapse prevention as usual
  Interventions: Behavioral: Discontinuity of care, non specialised care

INTERVENTIONS:
Behavioral: Continuity of specialized care — Continuity of care in treatment and professional caregiver was given during 5 year. Treatment targets included relapse prevention through recognition of prodromal symptoms, coping with negative symptoms and stress, increasing medication adherence, decrease of substance use, prevention of drop-out and stimulating and supporting participation in structural activities (work and/or education).
  Other Names: Relapse prevention; Specialized treatment; Maintenance antipsychotic medication
  Arms: Continuity of specialized care; Continuity of specialized care and parent groups
Behavioral: Parent groups combined with Continuity of Specialized care — Approximately fifty parent group therapy sessions will be held in a flexible way over a 60 month period. Each parent group was run by two experienced family therapists.
  Other Names: Family management as developed by Goldstein, Anderson, Falloon, Schooler and collaborators; Adaptation developed for parents of first psychotic episode patients as described in an earlier study of our group.
  Arms: Continuity of specialized care and parent groups
Behavioral: Discontinuity of care, non specialised care — Standard Treatment as usual (TU) was provided during 5 years by local mental health care professionals situated nearby the domicile of patients. TU had comparable treatment targets as ST but was not provided by treatment staff specialized in early intervention in schizophrenia or related disorders. However, TU was (like ST) sustained and dedicated to prevent psychotic relapse and improve social functioning.
  Other Names: Standard relapse prevention
  Arms: Treatment as usual

SUMMARY:
Objective: to evaluate the effectiveness of specialised and sustained intervention with or without parent groups during the initial phase of schizophrenia or related disorders on relapse prevention

Methods: A three conditions randomized trial with a duration of five years

Participants: 200 consecutively referred patients aged 15-28 years with a first psychotic episode of schizophrenia or related disorder

Treatment-conditions: Specialized Treatment of early schizophrenia (ST), ST including Parent groups (ST+P) and Treatment As Usual (TAU).

Outcome-measures: cumulative relapse rates and time to first relapse after first remission. Secondary outcome measure: social functioning.

Statistical analysis: cumulative relapse rates using life-table methods. The effect of the three interventions on time to first relapse after remission will be compared using Cox regression analysing intention to treat (ITT) grouping.

DETAILED DESCRIPTION:
Evidence for optimal duration and necessary ingredients of early and sustained specialized treatment from first episode psychosis till the end of the initial phase schizophrenia is still insufficient. Randomized trials with a treatment duration of six months to two years with favorable symptomatic and psychosocial results disappeared at five year follow-up. Other studies suggest that specialized treatment should last 5 years in order to be able to prevent instead of only delaying clinical and psychosocial deteriorating.

In this study we examine both the symptomatic (relapse) and psychosocial outcome of a three armed five year randomized trial in the initial phase of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible for the study if they: 1) met DSM-IV-Revised criteria for schizophrenia or related disorders, 2) were suffering from a first psychotic episode and 3) were living in contact with parent(s) or other relatives.

Exclusion Criteria:

* Patients with drug-related psychoses were not included.

Ages: 15 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 1997-09; Primary Completion 2007-02 (Actual); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in Psychotic relapse | at year 1, year 3 and year 5
  Participants will be followed for the duration of the 5 year outpatient treatment of the trial. During the trial the timing and number of psychotic relapses of each participant will be assessed using the Life Chart Schedule (LCS) at year 1, year 3 and year 5 after the start of the trial.
  Trained interviewers not involved in clinical treatment of patients will elicit with the LCS detailed information of symptoms, signs and treatment from respondents (patients and/or parents) and from clinical records. Respondents will be asked to indicate any changes in symptomatology since the last interview. All details will be fitted in a schedule with 6 months intervals.

SECONDARY OUTCOMES:
Change in Social functioning | at year 1, year 3 and year 5
  During the duration of the 5 year outpatient treatment of the trial social functioning of each participant will be assessed using the Life Chart Schedule (LCS) at year 1, year 3 and year 5 after the start of the trial.
  Detailed information of social functioning in work, study, school and relations will be elicited from respondents (patients and/or parents) and from clinical records. Respondents will be asked to indicate any changes in functioning since the last interview.All details will be fitted in a schedule with 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Don Linszen, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center University of Amsterdam, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Linszen D, Dingemans P, Lenior M. Early intervention and a five year follow up in young adults with a short duration of untreated psychosis: ethical implications. Schizophr Res. 2001 Aug 1;51(1):55-61. doi: 10.1016/s0920-9964(01)00239-0. PMID 11479066
- [Background] Linszen D, Lenior M, De Haan L, Dingemans P, Gersons B. Early intervention, untreated psychosis and the course of early schizophrenia. Br J Psychiatry Suppl. 1998;172(33):84-9. PMID 9764132
- [Background] Linszen D, Dingemans P, Van der Does JW, Nugter A, Scholte P, Lenior R, Goldstein MJ. Treatment, expressed emotion and relapse in recent onset schizophrenic disorders. Psychol Med. 1996 Mar;26(2):333-42. doi: 10.1017/s0033291700034723. PMID 8685289
- [Background] Lenior ME, Dingemans PM, Linszen DH, de Haan L, Schene AH. Social functioning and the course of early-onset schizophrenia: five-year follow-up of a psychosocial intervention. Br J Psychiatry. 2001 Jul;179:53-8. doi: 10.1192/bjp.179.1.53. PMID 11435269
- See also: The RAISE Early Treatment Program (ETP), led by John Kane, M.D., of the Feinstein Institute for Medical Research in Manhasset, NY, is conducting a similar RCT with the same population and a comparable design. — http://www.nimh.nih.gov/news/science-news/2011/nimh-raise-project-makes-progress-as-teams-refine-research-approaches.shtml